CLINICAL TRIAL: NCT04989322
Title: A Phase 2 Open-label Single-arm Study to Evaluate the Combination of Pembrolizumab, Lenvatinib and Chemotherapy in Non-small Cell Lung Cancer (NSCLC) Harbouring Targetable Mutation and Failed Standard Tyrosine Kinase Inhibitors
Brief Title: Pembrolizumab, Lenvatinib and Chemotherapy After TKIs in NSCLC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Dr Joanne CHIU (Other)
Responsible Party: Sponsor-Investigator, Dr Joanne CHIU, Assistant Professor, The University of Hong Kong
Organization: The University of Hong Kong (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 475-0708-MT-Lung; MK-3475-C50 (Other: MSD)
Record Dates: First submitted 2021-07-26; First posted 2021-08-04 (Actual); Last update posted 2021-12-08 (Actual); Status verified 2021-11

CONDITIONS: Nsclc; EGFR Activating Mutation; EGF-R Positive Non-Small Cell Lung Cancer; ALK Gene Rearrangement Positive; ROS1 Gene Rearrangement; ROS1 Positive NSCLC - Reactive Oxygen Species 1 Positive Non-Small Cell Lung Cancer
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — pembrolizumab; lenvatinib; Pemetrexed; Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Experimental)
  Interventions: Drug: Pembrolizumab; Drug: Lenvatinib; Drug: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: Pembrolizumab — 200 mg Q3W
Drug: Lenvatinib — 8 mg daily
Drug: Pemetrexed — 500 mg/m2 Q3W
Drug: Carboplatin — AUC5 Q3W

SUMMARY:
Adding chemotherapy or anti-VEGF to immunotherapy is an emerging strategy to enhance the efficacy of immunotherapy in many cancers. This phase 2 study aims to explore the preliminary efficacy of combination pembrolizumab with lenvatinib and chemotherapy in NSCLC patients with sensitizing EGFR, ALK, or ROS1 genetic aberration refractory to standard targeted therapy.

ELIGIBILITY:
Main Inclusion Criteria:

* Histologically proven NSCLC
* Unresectable or metastatic NSCLC, including squamous cell carcinoma, harboring sensitizing EGFR, ALK, or ROS1 genetic aberrations who have received standard of care targeted therapy and have progressed on treatment. Patients with known T790M mutation should have received osimertinib and failed.
* Measurable disease per RECIST 1.1
* ECOG performance status ≤ 1
* Adequate organ function
* Adequately controlled blood pressure

Main Exclusion Criteria:

* Prior exposure to immunotherapy or chemotherapy
* Active untreated brain metastasis and/or carcinomatous meningitis
* Active, known or suspected autoimmune disease
* History of (noninfectious) pneumonitis that required systemic steroids or current pneumonitis/interstitial lung disease
* Condition requiring systemic treatment with either corticosteroids (> 10 mg daily prednisone equivalent) or other immunosuppressive medications
* Baseline proteinuria ≥ 1 g/24 hrs
* Electrolyte abnormalities that have not been corrected
* Significant cardiovascular impairment
* Gastrointestinal pathology that might affect the absorption of lenvatinib
* Preexisting grade ≥ 3 gastrointestinal or non gastrointestinal fistula
* Bleeding or thrombotic disorders or subjects at risk for severe hemorrhage
* Radiographic evidence of intratumoral caviations, encasement, or invasion of a major blood vessel
* Known history of tuberculosis
* Active, acute, or chronic clinically significant infections requiring therapy, including hepatitis B, hepatitis C, and HIV
* ECG with long QTc interval ≥ 470 ms

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Estimated)
Dates: Start 2021-10-05 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Overall response rate | 24 months
  Proportion of patients who have a confirmed CR or PR per RECIST 1.1

SECONDARY OUTCOMES:
Progression-free survival | 24 months
  Time from randomization to the first documented disease progression per RECIST 1.1 or death due to any cause, whichever occurs first
Overall survival | 36 months
  Time from randomization to death from any cause or last follow-up date
The incidence, severity as graded by NCI CTCAE v5.0, seriousness and relationship to study medication of adverse events (AEs) | 24 months
  Safety and tolerability

CONTACTS AND LOCATIONS:
Locations (1):
- Queen Mary Hospital, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Chan HW, Tse CCL, Li YC, Leung R, Kwok GW, Wong JSL, Li KH, Tsang JWY, Li CW, Lo JWY, Tang V, Hui R, Yau T, Ho JCM, Chiu JWY. A phase 2, open-label, single-arm study evaluating the combination of pembrolizumab, lenvatinib, carboplatin and pemetrexed in patients with metastatic non-small cell lung cancer harbouring targetable genomic alterations who progressed on standard tyrosine kinase inhibitors. Invest New Drugs. 2025 Dec;43(6):1191-1200. doi: 10.1007/s10637-025-01589-6. Epub 2025 Nov 10. PMID 41212380